CLINICAL TRIAL: NCT04552626
Title: Acute Effects From Prolonged Inactivity and Physical Activity Interventions on Cortical Blood Flow and Arterials Stiffness in School-aged Adolescents.
Brief Title: Activity Breaks for Brain Health in Adolescents
Acronym: ABBaH teens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Swedish School of Sport and Health Sciences (Other)
Collaborators: The Knowledge Foundation (Unknown); IKEA (Unknown); Skandia (Unknown); Konsumentföreningen Stockholm (Unknown); Generation PEP (Unknown); COOP (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: Dnr 2020-02597
Record Dates: First submitted 2020-09-10; First posted 2020-09-17 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Healthy Adolescents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Prolonged sitting (social breaks) (Experimental)
  Interventions: Behavioral: Prolonged sitting (social breaks)
- Prolonged sitting with step-up exercise break (Experimental)
  Interventions: Behavioral: Prolonged sitting with step-up exercise break
- Prolonged sitting with simple resistance activity breaks (Experimental)
  Interventions: Behavioral: Prolonged sitting with simple resistance activity breaks

INTERVENTIONS:
Behavioral: Prolonged sitting (social breaks) — Participants are required to sit for 80 minutes doing schoolwork, with a toilet break in between. Every twenty minutes participants will have a short social break. Test day begins at 8:00 with pretest measures, followed by the intervention at about 9:00, which will end around 12:00, with subsequent posttest measures.
  Arms: Prolonged sitting (social breaks)
Behavioral: Prolonged sitting with step-up exercise break — Participants are required to sit for 80 minutes doing schoolwork, with a toilet break in between. Every twenty minutes participants will have a physical activity break, where they will perform a simple moderate-intensity step-up exercise for three minutes at a predetermined pace. Test day begins at 8:00 with pretest measures, followed by the intervention at about 9:30, which will end around 12:00, with subsequent posttest measures.
  Arms: Prolonged sitting with step-up exercise break
Behavioral: Prolonged sitting with simple resistance activity breaks — Participants are required to sit for 80 minutes doing schoolwork, with a toilet break in between. Every twenty minutes participants will have a physical activity break, where they will perform simple resistance activities following a video for about three minutes. Test day begins at 8:00 with pretest measures, followed by the intervention at about 9:30, which will end around 12:00, with subsequent posttest measures.
  Arms: Prolonged sitting with simple resistance activity breaks

SUMMARY:
The main aim for this study is to investigate to what extent physical activity of moderate or low intensity, relative to prolonged inactivity, may acutely alter neural activity-related prefrontal cortex oxygenated hemoglobin during a cognitive demanding task in 13- 15 year-old adolescents. The study is primarily focused on investigating these effects in ecologically valid conditions, i.e. activity patterns that closely resemble a typical day in school and using activity modes that are suitable in a school setting.

DETAILED DESCRIPTION:
The study will be a controlled crossover experimental trial with three conditions. Each participant will complete each of the three experimental conditions, separated by a washout period of minimum four days. Physical activity behaviours and sleep will be monitored the day/night before each test day. The first visit will be a familiarization session for the collection of demographic data, fitness testing, and acquaintance with experimental procedures. On the second, third, and fourth visits, participants will undergo three different standardized 80-minutes interventions in a randomized order. Before and immediately after the 80-minutes interventions, blood pressure, augmentation index, and cerebral hemodynamic response of the prefrontal cortex during standardized cognitive tasks (nback test) will be measured. Additionally, saliva samples will be collected the morning of the test day, and before and after the interventions.

ELIGIBILITY:
Exclusion Criteria:

* Ongoing medication that can affect central circulation or brain circulation
* Ongoing infection
* Inability to apprehend information about the study or to perform the tests

Ages: 13 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2020-12-16 (Actual); Study Completion 2020-12-16 (Actual)

PRIMARY OUTCOMES:
Changes in cerebral blood flow | before to after 80 minutes intervention
  Oxygenated and deoxygenated hemoglobin concentration changes measured with functional near-infrared spectroscopy

SECONDARY OUTCOMES:
Cognitive performance | before and after 80 minutes intervention
  nback cognitive test (time and accuracy)
Augmentation index | before and after 80 minutes intervention
  measure of arterial stiffness
Cortisol | morning; before and after 80 minutes intervention
  measured from saliva
Mood | at the beginning of the day; before and after 80 minutes intervention
  Positive and Negative Affect Schedule (PANAS) comprised of 20 affect states (10 positive and 10 negative), each affect state scored on a scale going from 1 (very slightly or not at all) to 5 (extremely)
Sleepiness | at the beginning of the day; before and after 80 minutes intervention
  Karolinska Sleepiness Questionnaire; goes from 1 (extremely alert) to 9 (extremely sleepy)
Alertness | at the beginning of the day; before and after 80 minutes intervention
  100mm Visual Analogue Scale (VAS); range: 'not at all' to 'completely alert'

CONTACTS AND LOCATIONS:
Overall Officials: Örjan Ekblom, PhD, Principal Investigator — The Swedish School of Sport and Health Sciences
Locations (1):
- The Swedish School of Sport and Health Sciences (GIH), Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kjellenberg K, Ekblom O, Tarassova O, Fernstrom M, Nyberg G, Ekblom MM, Helgadottir B, Heiland EG. Short, frequent physical activity breaks improve working memory while preserving cerebral blood flow in adolescents during prolonged sitting - AbbaH teen, a randomized crossover trial. BMC Public Health. 2024 Aug 2;24(1):2090. doi: 10.1186/s12889-024-19306-y. PMID 39095724
- [Derived] Heiland EG, Kjellenberg K, Tarassova O, Fernstrom M, Nyberg G, Ekblom MM, Helgadottir B, Ekblom O. ABBaH teens: Activity Breaks for Brain Health in adolescents: study protocol for a randomized crossover trial. Trials. 2022 Jan 6;23(1):22. doi: 10.1186/s13063-021-05972-5. PMID 34991692